CLINICAL TRIAL: NCT02056262
Title: Prevalence and Identification of Pathogenic Species and Genotypes of Bacterial Diversity in Relation to the Severity of Dental Caries
Brief Title: Pathogenic Species and Genotypes of Bacterial Diversity in Relation to the Severity of Dental Caries
Acronym: Caries Species
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: AOI/2012/LH; 2013-A01213-42 (Other: RCB number)
Record Dates: First submitted 2014-02-04; First posted 2014-02-05 (Estimated); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Dental Cavity
Keywords: Bacteria; microbial community; hygiene
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plaque and saliva samples; DNA analysis is aimed at describing microbial communities.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 3 to 16 years of age: Volunteers of 3 to 16 years of age, coming in to the hospital for a dental consultation. See inclusion/exclusion criteria.
  Intervention: Dental cavity evaluation Intervention: Saliva sampling Intervention: Plaque sampling
  Interventions: Other: Dental cavity evaluation; Biological: Saliva sampling; Biological: Plaque sampling
- 17 - 45 years of age: Volunteers of 17 to 45 years of age, coming in to the hospital for a dental consultation. See inclusion/exclusion criteria.
  Intervention: Dental cavity evaluation Intervention: Saliva sampling Intervention: Plaque sampling
  Interventions: Other: Dental cavity evaluation; Biological: Saliva sampling; Biological: Plaque sampling

INTERVENTIONS:
Other: Dental cavity evaluation — The dental cavities present will be evaluated using the ICDAS (International Caries Detection and Assessment System).
Biological: Saliva sampling — A saliva sample will be harvested.
Biological: Plaque sampling — Plaque samples from a healthy tooth and a tooth with a cavity will be harvested.

SUMMARY:
The primary objective of this study is to estimate the distribution of pathogenic species and genotypes of bacterial diversity in 7 stages ICDAS (International Caries Detection and Assessment System) corresponding to the severity of dental caries among patients aged 3-45 years consulting in the Dentistry Departments of the Nîmes University Hospital and the Montpellier University Hospital.

DETAILED DESCRIPTION:
Secondary objectives include:

* Compare the distribution of bacterial species in relation to stages of severity of caries
* Compare the results from plaque with those of saliva samples.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers aged 3 to 45 who come in to the hospital for a dental consultation
* Minors must have parental permission
* The patient must have given his/her informed and signed consent

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is pregnant, or breastfeeding
* The patient has been on antibiotics within the past two months
* Smokers
* Teeth under current care
* Parodontopathy
* Use of a mouthwash within the last week
* Insufficient numbers of healthy and/or teeth with carious lesions for carrying out the study

Ages: 3 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Volunteers aged 3 to 45 who come in to the hospital for a dental consultation.
  Patients are recruted according to age in order to form two groups: 1/2 of participants will be between 3 and 16 years of age; the other half of participants will be between 17 and 45 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2017-03-08 (Actual); Study Completion 2017-03-08 (Actual)

PRIMARY OUTCOMES:
Bacterial profile | Baseline (day 0)
  Bacterial profiles will be constructed using saliva and plaque samples.
ICDAS assessment | Baseline (day 0)
  Dental caries will be assessed using the ICDAS (International Caries Detection and Assessment System) system

SECONDARY OUTCOMES:
Studies were stopped during high school? yes/no | baseline (Day 0)
Does the patient have at least five fillings? yes/no | Baseline (day 0)
Does the patient have at least one filling and one missing tooth on the anterior sector following the carious lesion? yes/no | baseline (day 0)
Within the last 12 months, the patient has had dental care or tooth removal following the carious lesion? yes/no | baseline (day 0)
Yesterday, did the patient eat at least three snacks (or sugary or carbonated drinks) between meals? yes/no | Baseline (day 0)
Yesterday, did the patient brush his/her teeth fewer than 2 times? yes/no | baseline (day 0)
The patient has at least one carious lesion restricted to the enamel? yes/no | baseline (day 0)
The patient has at least one carious lesion restricted to the enamel on an anterior tooth or involving the smooth surface on a posterior tooth (yes/no) | baseline (day 0)
The patient has at least one carious lesion attacking the dentin or pulp. yes/no | baseline (day 0)
The patient has at least one carious lesion reaching dentin or pulp on an anterior tooth or on the smooth surface of a posterior tooth (yes/no) | baseline (day 0)

OTHER OUTCOMES:
Profession (or parents' professions) | baseline (day 0)
Age | baseline (day 0)
Sex | baseline (day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Hervé Léon, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (3):
- France (3):
  - CHRU de Montpellier - Centre de Soins, d'Enseignement et de Recherche Dentaires, Montpellier
  - CHRU de Montpellier - Hôpital La Colombière, Montpellier
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes